CLINICAL TRIAL: NCT02875847
Title: The Effects of Human Milk Oligosaccharides on Faecal Microbiota, Gastrointestinal Symptoms, Mucosal Immunity and Barrier Function in Irritable Bowel Syndrome: a Parellell, Double-blind, Randomised, Placebo-controlled Study
Brief Title: Effects of HMOs on Faecal Microbiota, Gastrointestinal Symptoms, Mucosal Immunity and Barrier Function in IBS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glycom A/S (Industry)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NATRIBS; Dnr: 548-16 (Other: Regionala Etikprövningsnämnden i Göteborg)
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HMO1 (Active Comparator): Daily bolus of HMO1
  Interventions: Dietary Supplement: HMO1
- HMO2 (Active Comparator): Daily bolus of HMO2
  Interventions: Dietary Supplement: HMO2
- Dextropur (Placebo Comparator): Daily bolus of dextropur
  Interventions: Dietary Supplement: Dextropur

INTERVENTIONS:
Dietary Supplement: HMO1
  Arms: HMO1
Dietary Supplement: HMO2
  Arms: HMO2
Dietary Supplement: Dextropur
  Arms: Dextropur

SUMMARY:
The study is a randomised, placebo-controlled, double-blind parallel study in IBS patients. A total of 60 adult patients diagnosed with IBS-C, -D or -A/M according to Rome IV criteria will be included. The participants will be randomized into one of three groups consuming either HMO (two groups) or placebo (one group).

The primary objective of the study is to establish the effect of HMOs on the faecal microbiota in IBS patients. Secondary objectives are to assess the effect on gastrointestinal symptoms, mucosal immunity, gut barrier function, quality of life, and anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Age between 18 and 75 years at visit 2
3. Fulfills definition of IBS-D, IBS-C or IBS-A/M according to Rome IV criteria
4. Have a global IBS-SSS score of >174 during the 2 weeks run-in period
5. Read, speak and understand Swedish
6. Ability and willingness to understand and comply with the study procedures

Exclusion Criteria:

1. Participation in a clinical intervention trial one month prior to screening visit and throughout the study.
2. Any known gastrointestinal disease(s) that may cause symptoms or may interfere with the trial outcome, as judged by the investigator; in particular

   * lactose intolerance
   * coeliac disease
3. Other severe disease(s) such as malignancy, diabetes, severe coronary disease, kidney disease or neurological disease, as judged by the investigator.
4. Severe psychiatric disease and/or psychological disturbance, as judged by the investigator.
5. Use of highly dosed probiotic supplements (yoghurt allowed) one month prior to the study and throughout the study. Excluded products are (i) probiotic supplements in the form of capsules, tablets, and powders in sachets, and (ii) probiotic food and drink products which contain high doses of probiotics. The excluded food and drink products are available in the form of yoghurts, drinking yoghurts, shots and drinks under brands such as Proviva, Actimel, Activia, Wellness, and Verum.
6. Consumption of antibiotic drugs one month prior to screening and throughout the study. Antibiotic use within the last three months prior to screening will be registered.
7. Consumption on a regular basis of medication that might interfere with symptom evaluation (as judged by the investigator) two weeks prior to screening and throughout the study. Specifically excluded drugs are opioids, NSAIDs on a weekly basis, regular use of laxatives and anti-diarrhoeal drugs, any drugs indicated for IBS symptoms.
8. Diagnosed with and treated for IBS for more than 10 years
9. Pregnant or lactating or wish to become pregnant during the period of the study.
10. Lack of suitability for participation in the study for any reason as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in intestinal bifidobacteria abundance | Baseline and after 4 weeks of intake

SECONDARY OUTCOMES:
Change from baseline of faecal microbiota profile | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of IBS symptoms as measured via the total score on the IBS Symptoms Severity Scale (IBS-SSS) and the proportion of responders in all patients and subgroup of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of intensity of abdominal pain and number of days of abdominal pain as measured on the 11 point Numeric Rating Scale (NRS-11) in all patients and subgroups of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of bowel habits as measured via the IBS-SSS, the Bristol Stool Form Scale (BSFS) and a bowel movement diary in all patients and subgroup of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of abdominal distention as measured via the IBS-SSS in all patients and subgroups of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of gastrointestinal symptoms as measured by the Gastrointestinal Symptom Rating Scale for IBS patients (GSRS-IBS) in all patients and subgroup of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of quality of life in IBS patients as measured by the IBS-QOL in all patients and subgroups of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of anxiety and depression as measured by the Hospital Anxiety and Depression Scales (HADS) in all patients and subgroups of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of gastrointestinal symptom specific anxiety as measured by the Visceral Sensitivity Index (VSI) in all patients and subgroup of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of severity of somatic symptoms as measured by the Patient Health Questionnaire-15 (PHQ-15) in all patients and subgroup of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of biomarkers of inflammation in all patients and subgroups of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of biomarkers of gut barrier function in all patients and subgroups of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out
Change from baseline of biomarkers of the gut-brain axis in all patients and subgroups of patients | Baseline and after 4 weeks of intake, and after 4 weeks of wash-out

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, MD, PhD, Principal Investigator — Department of Internal Medicine; Hans Törnblom, MD, PhD, Principal Investigator — Department of Internal Medicine; Lena Öhman, PhD, Principal Investigator — Department of Internal Medicine
Locations (1):
- SU Sahlgrenska, Department of Internal Medicine, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iribarren C, Tornblom H, Aziz I, Magnusson MK, Sundin J, Vigsnaes LK, Amundsen ID, McConnell B, Seitzberg D, Ohman L, Simren M. Human milk oligosaccharide supplementation in irritable bowel syndrome patients: A parallel, randomized, double-blind, placebo-controlled study. Neurogastroenterol Motil. 2020 Oct;32(10):e13920. doi: 10.1111/nmo.13920. Epub 2020 Jun 14. PMID 32536023